CLINICAL TRIAL: NCT04181398
Title: Low Grade Inflammation in Childhood Obesity : an Independent Risk Factor for Endothelial Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Inge Gies, Professor, Universitair Ziekenhuis Brussel
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Palomino
Record Dates: First submitted 2019-08-08; First posted 2019-11-29 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Obesity, Childhood; Obesity; Endothelial Dysfunction; Cardiovascular Risk Factor; Inflammation
MeSH Terms: conditions — Pediatric Obesity; Obesity; Inflammation | interventions — Anthropometry; Blood Pressure; Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Observational cohort study without blinding or randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline high hs-CRP (Experimental): Anthropometry:
  * Actual Height and weight
  * Calculated BMI from measured weight and height.
  * Pubertal development (Tanner stage)
  * Waist circumference
  * Skin fold measurement (Triceps and Subscapular)
  * Waist-to-height ratio.
  Blood pressure (mean of 3 measurements)
  Peripheral arterial tonometry
  Questionnaire
  Blood sample (hsCRP)
  Interventions: Diagnostic Test: Anthropometry; Diagnostic Test: Blood pressure; Diagnostic Test: Peripheral arterial tonometry; Other: Questionnaire; Diagnostic Test: Blood sample
- Baseline low hs-CRP (Experimental): Anthropometry:
  * Actual Height and weight
  * Calculated BMI from measured weight and height.
  * Pubertal development (Tanner stage)
  * Waist circumference
  * Skin fold measurement (Triceps and Subscapular)
  * Waist-to-height ratio.
  Blood pressure (mean of 3 measurements)
  Peripheral arterial tonometry
  Questionnaire
  Blood sample (hsCRP)
  Interventions: Diagnostic Test: Anthropometry; Diagnostic Test: Blood pressure; Diagnostic Test: Peripheral arterial tonometry; Other: Questionnaire; Diagnostic Test: Blood sample

INTERVENTIONS:
Diagnostic Test: Anthropometry — * Actual Height and weight
  * Calculated BMI from measured weight and height.
  * Pubertal development (Tanner stage)
  * Waist circumference
  * Skin fold measurement (Triceps and Subscapular)
  * Waist-to-height ratio will be calculated from measured height and waist circumference.
Diagnostic Test: Blood pressure — Blood pressure will be measured using an oscillometric, electronic device (Mindray). The blood pressure will be measured 3 times; the first measurement will not be taken into account and the mean of the second and third measurement will be considered as the real blood pressure.
Diagnostic Test: Peripheral arterial tonometry — The investigator will measure the pulse wave amplitude by using a finger plethysmograph (peripheral arterial tonometry). The investigator will use the EndoPAT device from Itamar Medical Ltd. At the end of the examination, the participants will be asked to give a VAS-score (Visual Analogue Pain scale).
Other: Questionnaire — General questionnaire on cardiovascular risk factors
Diagnostic Test: Blood sample — Blood sample for hs-CRP

SUMMARY:
Eligible candidates will be recruited within the children with overweight and obesity having a metabolic risk evaluation before treatment in the period 2006 and 2010 at the pediatric clinic of the UZ Brussel In total 60 participants will be investigated. Firstly, 30 participating patients with initially elevated hsCRP will be selected at random ( following the date of their initial investigation) and afterwards matched for age, BMI z-score, and blood pressure with the same number of patients without initially elevated hCRP values

Data will be collected as follows:

* questionnaires
* clinical examination/ anthropometry
* blood sample (hsCRP)
* peripheral arterial tonometry (endoPAT)

DETAILED DESCRIPTION:
Obesity and overweight have become an important health burden in children and adolescents, with 19% of all children between 5 and 18 years being either obese or overweight in Belgium. Obesity and especially visceral adiposity early in life may contribute to the development of cardiovascular disease at older age, as it shows tracking into adulthood and is be associated with cardiovascular risk factors such as dyslipidemia, insulin resistance, arterial hypertension and low grade inflammation, in a variable percentage.

Low grade inflammation, as assessed by hSCRP, was found to be present in 20.6 % and 19.8 % of overweight children and adolescents. In adults, hSCRP levels between 1 and 3 mg/L and above 3 mg/L are considered coronary disease risk factors.

Endothelial dysfunction, know to precede the formation of atherosclerotic plaque, can be assessed in a non-invasive manner in children by peripheral artery tonometry. Only few studies have been performed in obese children with this bed-side technique, showing either normal of a disturbed function, reflected by a lower reactive hyperemia index. The association with low grade inflammation however was assessed in only one study. The investigators hypothesize that in adolescents and young adults with a history of childhood obesity a more disturbed endothelial function will be present in those with and /or current elevated hSCRP value.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-21 years at the moment of evaluation
* BMI > 1.3 Standard Deviation Score at the initial evaluation
* Hs-CRP available at initial evaluation

Exclusion Criteria:

* Acute of chronic Infection at the time of the study visit
* Be or have been a smoker of tabacco

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Endothelial cell function | through study completion, an average of 1 year (measured once)
  Reactive hyperemia index (RHI) measured by the EndoPAT device.

SECONDARY OUTCOMES:
hs CRP level | through study completion, an average of 1 year (measured once)
  The investigators also hypothesized that low grade inflammation, and thus a rise in hs-CRP, will be persistent overtime.
BMI z-score | through study completion, an average of 1 year (measured once)
  The researchers want to investigate the evolution of the level of the obesity of the participants over time
Fat percentage by skin fold measurements | through study completion, an average of 1 year (measured once)
  The researchers want to investigate the evolution of the level of the obesity of the participants over time

CONTACTS AND LOCATIONS:
Overall Officials: Jean De Schepper, PhD, Principal Investigator — Universitair Ziekenhuis Brussel; Inge Gies, PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- University Hospital of Brussels, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT04181398/Prot_SAP_000.pdf